CLINICAL TRIAL: NCT00107640
Title: Costs of Preventing Alcohol Problems in Older Adults
Brief Title: Project SHARE (Senior Health and Alcohol Risk Education)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Susan Ettner, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NIAAATAL13990; R01AA013990 (NIH); 5R01AA013990-02 (NIH)
Record Dates: First submitted 2005-04-06; First posted 2005-04-07 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2010-09

CONDITIONS: Alcohol Consumption
Keywords: At-risk drinking; Alcohol education; Effectiveness; Cost-effectiveness
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients not assigned to the experimental condition received usual care, which may or may not have included alcohol education.
- Patient-provider education (Experimental): Experimental patients received an intervention consisting of the following components: written reports and educational materials, a telephone health educator intervention (at baseline, 3 and 6 months), and a brief provider intervention.
  Interventions: Behavioral: Patient-provider education

INTERVENTIONS:
Behavioral: Patient-provider education — Experimental patients received an intervention consisting of the following components: written reports and educational materials, a telephone health educator intervention (at baseline, 3 and 6 months), and a brief provider intervention.
  Arms: Patient-provider education

SUMMARY:
Older adults become more sensitive to alcohol, and alcohol also interacts adversely with their common medical conditions and medications. The aim of Project SHARE (Senior Health and Alcohol Risk Education) is to see whether patient and provider education can decrease risky alcohol use and reduce health care costs in persons 60 years of age and older.

DETAILED DESCRIPTION:
Alcohol use in the elderly is an increasingly important public health problem. Alcohol-related risks and problems in older persons may come from the interaction between alcohol and diminished health or medication use. The proposed study is a randomized trial of the effectiveness and cost-effectiveness of an integrated patient-provider intervention to prevent risky alcohol use among older adults. The intervention will include a tested screening and education system that was developed especially for older adults and their providers, supplemented by a well-established intervention for physicians. The proposed research design involves randomization of 31 primary care physicians in seven clinics and their eligible patients aged 60+ to the intervention versus "usual care."

ELIGIBILITY:
Inclusion Criteria:

* 60 and over
* At-risk drinkers
* Patient of participating physician

Exclusion Criteria:

* Severe cognitive impairment
* Terminally ill or deceased
* Expected to move out of area or into nursing home within following year
* Could not fill out written surveys in English
* Likely dependent drinker

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2005-05; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
At-risk drinking at 6 month followup | 6 months
  At-risk drinking is alcohol use that (either alone or in conjunction with selected comorbidities, symptoms and/or medications) poses health risks. It is measured using the CARET instrument developed by Moore and colleagues.
At-risk drinking at 12 month followup | 12 months
  At-risk drinking is alcohol use that (either alone or in conjunction with selected comorbidities, symptoms and/or medications) poses health risks. It is measured using the CARET instrument developed by Moore and colleagues.

SECONDARY OUTCOMES:
Health-related quality of life at 6 months | 6 months
  Health-related quality of life (HRQL) is measured using the SF-6D.
Depressive symptoms | 12 months
  Depressive symptoms are measured using the Geriatric Depression Scale.
Mental Composite Score at 6 months | 6 months
  We used self-reported SF12 data from baseline, 6- and 12-month written surveys to construct Mental Composite Score (MCS) and Physical Composite Score (PCS).
Healthcare utilization | 12 months (cumulative)
  We used self-reported data from 3-month, 6-month and 12-month written patient surveys to measure cumulative healthcare utilization by type (e.g., hospitalizations, emergency department visits, physician visits, etc.) over the twelve months following baseline.
Outpatient service costs | 12 months (cumulative)
  We used administrative data on clinic-based services linked to Medicare fee schedules to construct cumulative measures of outpatient service costs (from the Medicare perspective) for the twelve months following baseline.
Direct recruitment and intervention costs | 12 months (cumulative)
  We collected data on the resources used directly for recruitment (e.g., clinic-based staff time, phones, postage, etc.) and the intervention (e.g., cost of health educator time, supplies, opportunity costs of the physician's time, etc.) spent on the intervention, to construct overall measures of the per-patient cost of recruitment and intervention.
Health-related quality of life at 12 month followup | 12 months
  Health-related quality of life (HRQL) is measured using the SF-6D.
Mental Composite Score at 12 month followup | 12 months
  We used self-reported SF12 data from baseline, 6- and 12-month written surveys to construct Mental Composite Score (MCS) and Physical Composite Score (PCS).
Physical Composite Score at 6 month followup | 6 months
  We used self-reported SF12 data from baseline, 6- and 12-month written surveys to construct Mental Composite Score (MCS) and Physical Composite Score (PCS).
Physical Composite Score at 12 month followup | 12 months
  We used self-reported SF12 data from baseline, 6- and 12-month written surveys to construct Mental Composite Score (MCS) and Physical Composite Score (PCS).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Ettner, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Sansum-Santa Barbara Medical Foundation Clinics, Santa Barbara, California, United States

REFERENCES:
- [Derived] Barnes AJ, Xu H, Tseng CH, Ang A, Tallen L, Moore AA, Marshall DC, Mirkin M, Ransohoff K, Duru OK, Ettner SL. The Effect of a Patient-Provider Educational Intervention to Reduce At-Risk Drinking on Changes in Health and Health-Related Quality of Life Among Older Adults: The Project SHARE Study. J Subst Abuse Treat. 2016 Jan;60:14-20. doi: 10.1016/j.jsat.2015.06.019. Epub 2015 Jul 8. PMID 26254687
- [Derived] Ettner SL, Xu H, Duru OK, Ang A, Tseng CH, Tallen L, Barnes A, Mirkin M, Ransohoff K, Moore AA. The effect of an educational intervention on alcohol consumption, at-risk drinking, and health care utilization in older adults: the Project SHARE study. J Stud Alcohol Drugs. 2014 May;75(3):447-57. doi: 10.15288/jsad.2014.75.447. PMID 24766757
- See also: Sansum - Santa Barbara Medical Foundation Clinic — http://www.sansumclinic.org/